CLINICAL TRIAL: NCT04379687
Title: Immersive Virtual Reality in Post Stroke Physiotherapy
Brief Title: Immersive Virtual Reality in Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yolanda Marcen Roman (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Sponsor-Investigator, Yolanda Marcen Roman, Principal investigador, Instituto de Investigación Sanitaria Aragón
Organization: Instituto de Investigación Sanitaria Aragón (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VR stroke
Record Dates: First submitted 2020-04-17; First posted 2020-05-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Balance; Stroke; Physical Therapy; Virtual Reality
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): 1. st part: Conventional physiotherapy treatment program aimed at achieving functional improvement and increased postural control. 15 minutes
  2. nd part: Experimental training program for static and dynamic balance in sitting and standing by immersive Virtual Reality. 15 minutes
  Interventions: Other: Virtual reality
- Control group (Active Comparator): 1. st part: Conventional physiotherapy treatment program aimed at achieving functional improvement and increased postural control.15 minutes
  2. nd part: Training program for static and dynamic balance in sitting and standing, according to Bayouk. 15 minutes
  Interventions: Other: Control group

INTERVENTIONS:
Other: Virtual reality — Use of virtual reality glasses for balance work
  Arms: Virtual reality
Other: Control group — Balance treatment with according to Bayouk physiotherapy
  Arms: Control group

SUMMARY:
Physiotherapy intervention programs in the post-stroke patient should develop strategies to assess functional deficit, prevent poorly adaptive plasticity and maximize functional gain. For relearning and functional training, the required activities require motor control and must comply with the following principles: movements close to normal, muscular activation, movement conduction, focused attention, repetition of desired movements, specificity of training, intensity and transfer. These principles underlie the most widely used conventional physiotherapy intervention programs in the hospital setting.

Advances in technology have made it possible to start using immersive VR in the therapeutic approach to various pathologies that affect motor function.

DETAILED DESCRIPTION:
Physiotherapy intervention programs in the post-stroke patient should develop strategies to assess functional deficit, prevent poorly adaptive plasticity and maximize functional gain. For relearning and functional training, the required activities require motor control and must comply with the following principles: movements close to normal, muscular activation, movement conduction, focused attention, repetition of desired movements, specificity of training, intensity and transfer. These principles underlie the physiotherapy intervention programs specifically most used in the hospital setting.

Main aims

1-To determine if the designed immersive VR training program is better in the short term (15 sessions) and in the medium term (30 sessions) than the conventional physiotherapy training with respect to the change of the parameters related to the static balance in sitting and standing and dynamic balance in post-stroke patients.

Secondary aims 2. To determine the efficacy in the short term (15 sessions) and in the medium term (30 sessions) of immersive VR systems compared to conventional physiotherapy procedures regarding the quality of life associated with stroke, the degree of independence and autonomy .

3. To determine the safety of the application of training programs in immersive VR settings in post-stroke subjects with respect to the number of adverse effects produced.

4. Determine prognostic factors associated with insufficient improvement (less than moderate change) after stroke treatment with the designed immersive VR program and with conventional physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults> 18 years and <80 years.
* Diagnosis of hemiparesis or post-stroke hemiplegia.
* Minimum score of 2 points on item 3.2 of the Berg Scale, which establishes that the patient can remain in a sitting position for 30s without help.

Exclusion Criteria:

* Aphasia, scores over 45 on the Mississippi Aphasia Screening Test.
* Cerebellar pathology.
* Hemineglect or previous neurological disorder.
* Visual disturbances that prevent the use of VR glasses.
* Moderate cognitive decline, scores less than 43 on the Mini-mental State examination.
* Previous musculoskeletal disorders that make it difficult or impossible to balance sitting and standing or walking.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Postural Assessment Scale for Stroke Patients (PASS). | 45 minutes
  Static balance and functional mobility, This consists of 12 items and is subdivided into two parts: mobility (7 items) and balance (5 items), each with a score ranging from 0 (minimum) to 3 (maximum); the total scale score is 36 points.
  The PASS is made up of 12 items of increasing difficulty, of a 4-point scale in which items are scored from 0 to 3. The total score varies from 0 to 36
10 meter walk test. | 15 minutes
  Dynamic balance and gait
Berg Balance Scale | 15 minutes
  Static balance and functional mobility The Berg scale comprises 14 items (score comprised 0-4). Total scores can range from 0 (severely impaired balance) to 56 (excellent balance).
Balance Evaluation Systems Test (BESTtest) | 45 minutes
  Static balance and functional mobility
Timed Get uo and go test | 10 minutes
  Dynamic balance and gait

SECONDARY OUTCOMES:
Stroke-specific quality of life scale (ECVI-38) | 15 minutes
  Quality of life associated with stroke It has comprises 38 items, (score comprised 1-5). Total scores can range from 38 (excellent) to 190 point (very poor quality of life)
The Barthel Index | 10 minutes
  Degree of autonomy The sum of the scores obtained will determine the degree of dependency, so if the person is less than 20, they are considered totally dependent, if they are between 40 and 55, they are moderately dependent, if they are over 60, they are considered to be dependent mild and if it is 100 it will be totally independent (95 in case you need the use of a wheelchair
Ad hoc questionnaire | 10 minutes
  Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Aitor Garay Sanchez, Master, Study Chair — IIS Aragón; Mercedes Ferrando Margeli, Master, Principal Investigator — IIS Aragón; María Ángeles Franco Sierra, PhD, Principal Investigator — IIS Aragón
Locations (1):
- Hospital universitario Miguel servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grefkes C, Fink GR. Connectivity-based approaches in stroke and recovery of function. Lancet Neurol. 2014 Feb;13(2):206-16. doi: 10.1016/S1474-4422(13)70264-3. PMID 24457190
- [Background] Hugues A, Di Marco J, Janiaud P, Xue Y, Pires J, Khademi H, Cucherat M, Bonan I, Gueyffier F, Rode G. Efficiency of physical therapy on postural imbalance after stroke: study protocol for a systematic review and meta-analysis. BMJ Open. 2017 Jan 30;7(1):e013348. doi: 10.1136/bmjopen-2016-013348. PMID 28137928
- [Background] Freburger JK, Li D, Johnson AM, Fraher EP. Physical and Occupational Therapy From the Acute to Community Setting After Stroke: Predictors of Use, Continuity of Care, and Timeliness of Care. Arch Phys Med Rehabil. 2018 Jun;99(6):1077-1089.e7. doi: 10.1016/j.apmr.2017.03.007. Epub 2017 Apr 4. PMID 28389108
- [Background] Li S. Spasticity, Motor Recovery, and Neural Plasticity after Stroke. Front Neurol. 2017 Apr 3;8:120. doi: 10.3389/fneur.2017.00120. eCollection 2017. PMID 28421032
- [Background] Kim A, Darakjian N, Finley JM. Walking in fully immersive virtual environments: an evaluation of potential adverse effects in older adults and individuals with Parkinson's disease. J Neuroeng Rehabil. 2017 Feb 21;14(1):16. doi: 10.1186/s12984-017-0225-2. PMID 28222783
- [Background] Yasuda K, Muroi D, Ohira M, Iwata H. Validation of an immersive virtual reality system for training near and far space neglect in individuals with stroke: a pilot study. Top Stroke Rehabil. 2017 Oct;24(7):533-538. doi: 10.1080/10749357.2017.1351069. Epub 2017 Jul 12. PMID 28701101
- [Background] Llorens R, Noe E, Colomer C, Alcaniz M. Effectiveness, usability, and cost-benefit of a virtual reality-based telerehabilitation program for balance recovery after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2015 Mar;96(3):418-425.e2. doi: 10.1016/j.apmr.2014.10.019. Epub 2014 Nov 13. PMID 25448245
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493